CLINICAL TRIAL: NCT01072201
Title: To Access the Effects of Mucositis in Adults With Dental Implants
Acronym: implantitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRO-0107-PERIO-MUC-ITA-PC
Record Dates: First submitted 2008-09-26; First posted 2010-02-19 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Mucositis
MeSH Terms: conditions — Mucositis | interventions — Triclosan; Fluorides; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total toothpaste (Experimental): Triclosan/copolymer/fluoride toothpaste
  Interventions: Drug: Triclosan and Fluoride
- Ultrabrite toothpaste (Placebo Comparator): Fluoride Toothpaste
  Interventions: Drug: Fluoride

INTERVENTIONS:
Drug: Triclosan and Fluoride — Brush twice daily
  Other Names: Total Toothpaste
  Arms: Total toothpaste
Drug: Fluoride — Brush twice daily
  Other Names: Ultrabrite toothpaste
  Arms: Ultrabrite toothpaste

SUMMARY:
Clinical research for the treatment of mucositis subjects who have dental implants for a minimum of one-year.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 30-70.
* Availability for the six-month duration of the clinical research study.
* Good general health.
* Subjects who have lost teeth for periodontal disease reasons and who have been restored with implants.
* Minimum of 5 remaining teeth and a minimum of 2 implants.
* Initial evaluation of the gingival and peri-implant mucosal tissues by determining full mouth bleeding on probing.
* Initial plaque evaluation by determining full mouth presence/absence of plaque.
* Signed Informed Consent Form.

Exclusion Criteria:

* Tumor(s) of the soft or hard tissues of the oral cavity.
* Untreated periodontal disease (purulent exudate, tooth mobility, and/or extensive loss or periodontal attachment or alveolar bone).
* Carious lesions requiring immediate restorative treatment.
* Uncontrolled Diabetes
* Use of antibiotics any time during the one month prior to entry into the study.
* Untreated peri-implantitis.
* Participation in any other clinical research study or test panel within the three months prior to entry into the study.
* Pregnant women or women who are breast feeding.
* History of allergies to personal care/consumer products or their ingredients.
* Medical condition which prohibits not eating/drinking for up to 2 hours.
* Current alcohol or drug abuse.
* Systemic or local disease conditions that would compromise post-operative healing.
* Regular use of anti-inflammatory drugs.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Ramberg, DDS, Principal Investigator
Locations (1):
- Ariminum Research & Dental Education Center, Rimini, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Toothpaste: Triclosan/copolymer/Fluoride
- Ultrabrite Toothpaste: sodium fluoride control(placebo)
Period: Overall Study
Arm/Group | Total Toothpaste | Ultrabrite Toothpaste
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ultrabrite Toothpaste: sodium fluoride control (placebo)
- Total: Total of all reporting groups
Arm/Group | Total Toothpaste | Ultrabrite Toothpaste | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 52
  >=65 years | 4 | 4 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 57.36 (7.38) | 57.83 (7.97) | 57.59 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Bleeding on Probing
Description: Percentage of Bleeding Scale: The bleeding sites are identified by either a 0 or 1. (0=no bleeding & 1= bleeding) The number of spots between teeth that bleed are divided by number of spots between teeth that are scored.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage of bleeding sites
Arm/Group | Total Toothpaste | Ultrabrite Toothpaste
Number analyzed (Participants) | 30 | 29
Percentage of bleeding sites | 53.8 (17.6) | 52.3 (24.6)
Statistical Analysis 1: Comparison: Total Toothpaste vs Ultrabrite Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Mean Pocket Depth
Description: Measurement scale: 0 millimeter measurement= no pocket depth. 3, 4, 5, & 6 millimeter are indications of deeper Pocket depth.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Total Toothpaste | Ultrabrite Toothpaste
Number analyzed (Participants) | 30 | 29
Millimeters | 4.4 (0.6) | 4.5 (0.5)
Statistical Analysis 1: Comparison: Total Toothpaste vs Ultrabrite Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

3. Primary Outcome: Mean Percentage of Plaque Scores
Description: Mean Percentage (%) of dental plaque on all tooth surfaces, including implants and natural teeth. Plaque Scale is 0=no plaque and 1= dental plaque present. Percentage is derived from sum of all plaque scores divided by the number of tooth surfaces scored.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of dental plaque
Arm/Group | Total Toothpaste | Ultrabrite Toothpaste
Number analyzed (Participants) | 30 | 29
percentage of dental plaque | 13.2 (15.6) | 16.0 (17.8)
Statistical Analysis 1: Comparison: Total Toothpaste vs Ultrabrite Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | Total Toothpaste | Ultrabrite Toothpaste
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days